CLINICAL TRIAL: NCT02600585
Title: Post-Marketing Observational Study of Safety Following Vaccination With Flublok® Compared to Licensed IIV in Adults 18 Years of Age and Older
Brief Title: Post-Marketing Observational Study of Safety Following Vaccination With Flublok® Compared to Licensed IIV in Adults
Status: Completed | Type: Observational
Sponsor: Protein Sciences Corporation (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: PSC13
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Human Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Flublok: Recombinant influenza vaccine (RIV); Intramuscular injection of vaccine of recombinant uncleaved hemagglutinin (rHA0) derived from influenza A/H1N1, A/H3N2, and B viruses, as identified for the season by the FDA Vaccines and Related Biological Products Advisory Committee (VRBPAC) in a total volume of 0.5 mL.
  Interventions: Biological: Recombinant Influenza Vaccine
- Inactivated Influenza Vaccine: Injectable, inactivated, egg-based influenza vaccines (IIV); Intramuscular injection of vaccine (whether trivalent or quadrivalent) derived from influenza A/H1N1, A/H3N2, and B viruses, as identified for the season by the FDA Vaccines and Related Biological Products Advisory Committee (VRBPAC) in a total volume of 0.5 mL.
  Interventions: Biological: Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Recombinant Influenza Vaccine — Intramuscular injection of study vaccine
  Other Names: Flublok
  Groups: Flublok
Biological: Inactivated Influenza Vaccine — Intramuscular injection of study vaccine
  Groups: Inactivated Influenza Vaccine

SUMMARY:
The primary objective of this study is to retrospectively characterize the safety of Flublok in adults 18 years of age and older, in comparison with egg-based trivalent or quadrivalent inactivated influenza vaccines (IIVs), using a methodological approach designed to query the database of electronic health records (EHR) maintained by Kaiser-Permanente, Northern California (KPNC), a large medical care organization (MCO).

DETAILED DESCRIPTION:
The primary analysis is a nonrandomized, observational retrospective cohort study. Data on adults 18 years of age and older who were enrolled in the KPNC database during the risk intervals after vaccination analyzed for this study who were vaccinated with Flublok or an IIV (either IIV3 or IIV4) will be identified for analysis. The rates of occurrence of specific MAEs of interest in pre-specified risk intervals following Flublok and IIV will be compared.

ELIGIBILITY:
Inclusion Criteria:

Data from the EHR of all adult KPNC members 18 years of age and older, who received Flublok for active immunization against influenza as part of routine medical care within the KPNC system. The comparator cohort will include data from all adults in the same age group who received any IIV (trivalent or quadrivalent) during the period of Flublok administration.

Exclusion Criteria:

Healthcare providers are expected not to administer Flublok or IIV to individuals with known contraindication to either vaccine (see product package inserts). However, there will be no exclusions other than age and KPNC membership criteria at the time of vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adults 18 years of age and older who are vaccinated with either Flublok or IIV within the same time period, e.g. month of the year.
Sampling Method: Probability Sample
Enrollment: 254648 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious adverse events (SAEs) and medically-attended adverse events (MAEs) | Five months post-vaccination
  Incidence of Serious and/or Medically-Attended Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Roger Baxter, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Vaccine Study Center, Oakland, California, United States